CLINICAL TRIAL: NCT01816347
Title: Evaluation of Pre-deployment Device-to-artery Relative Axial Motion in Coronary Catheterizations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-61-11
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Routine PCI patients
  Interventions: Procedure: Routine PCI

INTERVENTIONS:
Procedure: Routine PCI

SUMMARY:
The cyclic movement of the heart and the coronary arteries induces relative axial movement between the artery and a pre-deployed intra-luminal stent which may cause malpositioning. Using a new imaging algorithm to indicate the position of a stent in patients undergoing percutaneous coronary intervention (PCI), the investigators will measure the pre-deployment relative, intra-luminal stent axial movement in the different coronary arteries to facilitate the precise deployment site.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine PCI

Exclusion Criteria:

* Unstable patients

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine PCI
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Relative axial movement of predeployed stent | One month

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel